CLINICAL TRIAL: NCT02395315
Title: Placement of Hydrophilic TiZr Implants to Enhance Implant Survival in Diabetic Patients: A Prospective, Two-arm, Cohort Study
Brief Title: Alveolar Bone Changes in Diabetes (ABCD) Study
Acronym: ABCD
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: Tamirshalev
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Osseointegration; Bone vascularity; Primary implant stability
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Well-controlled diabetic (WC): well-controlled diabetic controls (HbA1c ≤ 7.0%), individuals will receive a single 4.1 Titanium-Zirconia, hydrophilic (Roxolid) implant placed in the posterior mandible, a bone core will be taken for histologic and histomorphometric analysis.
  Interventions: Device: Well-controlled diabetic (WC)
- Poorly controlled diabetics (PC): Poorly controlled diabetics (HbA1c >7.5% & <10%), individuals will receive a single 4.1 Titanium-Zirconia, hydrophilic (Roxolid) implant placed in the posterior mandible, a bone core will be taken for histologic and histomorphometric analysis.
  Interventions: Device: Poorly controlled diabetics (PC)

INTERVENTIONS:
Device: Well-controlled diabetic (WC) — Each individual will receive one implant (4.1 Titanium-Zirconia, hydrophilic-Roxolid), that will be placed in the posterior mandible.
  Groups: Well-controlled diabetic (WC)
Device: Poorly controlled diabetics (PC) — Each individual will receive one implant (4.1 Titanium-Zirconia, hydrophilic-Roxolid), that will be placed in the posterior mandible.
  Groups: Poorly controlled diabetics (PC)

SUMMARY:
Type 2 Diabetes Mellitus (DM) is a very prevalent metabolic disorder in the adult population affecting roughly 17.7 million people in the US alone. The harmful effect of DM on implant integration and survival has been attributed to vascular complications in the alveolar bone that lead to compromised blood supply and decreased bone density. Nonetheless, the specific detrimental effects of DM in the alveolar bone have not been investigated in humans.

People with DM generally lose more teeth than persons without diabetes, but implant placement in not well controlled diabetics is not routinely performed due to the lack of relevant evidence and the risk for implant failure and associated complications. Chemically modified, micro-rough, hydrophilic (SLActive®) titanium implant surfaces have been shown to accelerate osseointegration of dental implants placed in diabetic animals. It has been hypothesized that this enhanced biologic response is due to the biocompatibility and hydrophilicity of the surface that actively attracts blood and is populated by progenitor cells, and growth factors that improve stromal cell differentiation.

Hypotheses:

It is hypothesized that hyperglycemia results in compromised vascularity in the mandible. Thus, hydrophilic TiZr implant surfaces (Roxolid®) that actively attract fluids and possess excellent osteoconductive properties, may enhance peri-implant bone response in diabetic patients to levels comparable to well-controlled diabetics.

DETAILED DESCRIPTION:
A high level of evidence exists to support the placement of implants in type 2 diabetics with glucosylated hemoglobin (HbA1c) levels within the normoglycemic range. Less information is available for the integration of implants placed in diabetics that cannot achieve good glycemic control, who may represent up to 50% of the diabetic patient population. Recent data from the medical literature have unveiled the deleterious effect of uncontrolled diabetes mellitus (DM) on the bone marrow. The microvascular alterations of DM on skeletal bones lead to microangiopathy, reduced blood flow and fatty degeneration in the bone marrow. Nascent theories that are founded upon the observation of increased levels of soluble osteoprotegerin (OPG) levels in uncontrolled DM implicate disruption of RANKL/OPG signaling as a potential pathway for the diabetes- related bone alterations. Nonetheless, no data is currently available on the pathophysiology of the alveolar bone in patients with DM.

It is hypothesized that 1) hyperglycemia results in compromised vascularity in the mandible, thus 2) hydrophilic TiZr implant surfaces (Roxolid®) that actively attract fluids and possess excellent osteoconductive properties, may enhance peri-implant bone response in not well-controlled diabetics (NCD) to levels comparable to well-controlled diabetics (WCD). We further hypothesize that the expected decreased RANKL/OPG ratio in NCD versus WCD will not recover during post-surgery bone remodeling. To assess our hypotheses, we will recruit n=21 type II WCD (HbA1c≤7.0%) and n=21 type II NCD (7.5%<HbA1c≤10%) seeking implant placement in the mandible. We will collect intra-operative bone specimens at baseline and blood samples to assess bone structural alterations (H&E stain), microvascular density (immunohistochemistry), bound RANKL/OPG (immunohistochemistry) and serum RANKL/OPG (ELISA). Implant integration and success will be assessed at 3, 6, 12 and 36-months.

Obtained results will give dental researchers new insights into the pathophysiology of the alveolar bone in diabetes and will provide information on the safety and efficacy of implant placement in type II diabetic patients that cannot control their glycemic status. Collectively, this work will pave the way for identifying efficacious implant treatment modalities for persons that live with type II diabetes to alleviate the morbidity associated with tooth loss in this susceptible population group.

ELIGIBILITY:
Inclusion Criteria:

Adult patients aged 18-85 years with diagnosed DM2.

History of DM2 for at least two years prior to enrollment.

At least one edentulous site in the canine or posterior mandible regions.

HbA1c >7.5% & <10% for enrollment in the test group.

HbA1c ≤ 7.0% for enrollment in the control group.

Available for follow up at 12 months.

Exclusion Criteria:

Mandibular incisor sites that will not allow bone core retrieval due to limited alveolar bone width (ridge width <5mm, height <10mm) as confirmed by pre-operative CBCT.

Smokers: current, or ex-smokers with <2 years cessation.

Active periodontal disease.

Medications that affect bone healing (e.g. bisphosphonates or chronic steroids).

Patients who are carriers of transmissible disease(s) that may unnecessarily expose laboratory personnel to risks.

Participants with a physician-diagnosed osteoporosis (Z-score ≤ -2).

Females during pregnancy or lactation and females that plan to become pregnant in the following year.

Patients that will not agree to participate in this study or sign the consent form.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosed type II DM exhibiting at least one edentulous site in the posterior mandible or canine region presenting with levels of HbA1c >7.5% & <10% for enrollment in the PC group and HbA1c ≤ 7.0% for enrollment in the WC group.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2021-11-07 (Actual)

PRIMARY OUTCOMES:
Differences in alveolar bone vascularity among well-controlled and not well-controlled diabetic patients. | Baseline (intra-operative bone sample)
  The difference between alveolar bone vascularity of well-controlled and not well-controlled diabetic patients by immunostaining

SECONDARY OUTCOMES:
RANK-L to OPG ratio | Baseline to 8 weeks
  A comparison between RANK-L to OPG ratio to determine the state of bone remodeling in each cohort.

OTHER OUTCOMES:
Differences in alveolar bone mineralization | Baseline (intra-operative bone sample)
  Comparison of bone mineralization between the two cohorts via histomorphometric measurement of vital bone percentage at the time of implant surgery
ISQ values as a surrogate for implant stability | Time of implant surgery-36 months
  Recording of the ISQ values (Osstel) and maximum insertion torque during implant placement as surrogates for primary implant stability.
Implant survival and success assessment at 3-months, 6-months, 1-year and 3-years post-loading | 3 years
  Implant survival and success assessment at 3-months, 6-months, 1-year and 3-years post-loading
Marginal bone level assessment | 3 years
  Assessment of marginal bone level maintenance around the implants at 3-months, 6-months, 1-year and 3-years post-loading. Periapical radiographs will be obtained using a paralleling technique with customized film holders will be obtained at baseline
Implant surgery-related complications | 3 months
  Short-term soft tissue and implant-related complications associated with implant surgery recorded at every post-op visit up to 3-months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: George Kotsakis, DDS, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - University of Minnesota Advanced Education in Periodontology, Minneapolis, Minnesota
  - University of Texas, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided